CLINICAL TRIAL: NCT04040842
Title: Quality and Outcomes in Global Cancer Surgery: a Prospective, International Cohort Study Evaluating Low Anterior Resection Syndrome (LARS)
Brief Title: International Low Anterior Resection Score Evaluation
Acronym: PrePostLARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: King's College London (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Audrius Dulskas, Assoc. professor, National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos
Other Study IDs: ISUCRS
Record Dates: First submitted 2019-07-28; First posted 2019-08-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Rectal cancer; low anterior resection; low anterior resection syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients undergoing low anterior resection — Patients before the surgery and one year after the surgery will be assessed with questionnaire.

SUMMARY:
* Aim: The aim of this study is to perform a prospective, international 4 months cohort study evaluating bowel function before curative rectal cancer surgery and one year after the surgery using the LARS score.
* Primary outcome measure: LARS score before surgery and 1 year after the surgery.
* Primary comparison: Between average LARS score before and after curative surgery and also comparing these with publish LARS score on normal population.

DETAILED DESCRIPTION:
All patients undergoing treatment for rectal rectal will be included in the study. Before any treatment all the included patients will be asked to fill the LARS score (5 question questionnaire with differently weighted answers for assessing the low anterior resection score). One year after the low anterior resection (without the stoma) or following the stoma take down patients will be reassessed. The LARS score will be filled one again. Patient characteristics, age, cancer stage, level of anastomosis will be assessed aswel.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing rectal cancer surgery on curative intent.
* Elective surgery patients.
* Laparoscopic, laparoscopic-converted, robotic, TaTME (transanal total mesorectal excision) and open cases will be included.
* Patients aged 18 years and over should be included.

Exclusion Criteria:

* Patients undergoing a procedure purely for diagnosis or staging should be excluded.
* Patients with palliative treatment.
* Patients with recurrence should be excluded.
* Patients with dementia
* Patients who do not complete their treatment within 12 months of primary surgery e.g. including reversal of stoma, chemotherapy etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to perform a prospective, international 4 months cohort study evaluating bowel function before curative rectal cancer surgery and one year after the surgery using the LARS score.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
LARS score change comparing before surgery and 1 year after the surgery. | 12 months
  Low anterior resection score is a simple questionnaire consisting of five simple questions for bowel function assessment after anterior resection. The maximum number is between 0 and 42. No LARS (good bowel function) is from 0 to 20; minor LARS - 21-29 and major LARS (poor bowel function) more than 29.
  Between average LARS score before and after curative surgery and also comparing these with published LARS score on normal population.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Nunoo-Mensah, MD, Study Director — King's College
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided